CLINICAL TRIAL: NCT01614678
Title: AIR OPTIX® COLORS: Automated vs Semi-automated Manufacturing Processes
Brief Title: A Comparison of Manufacturing Processes for AIR OPTIX® COLORS Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: P-383-C-005/C-12-026; C-12-026 (Other: Alcon)
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2014-02

CONDITIONS: Myopia
Keywords: myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX® COLORS Auto, then AIR OPTIX® COLORS Semi-auto (Other): Lotrafilcon B contact lens with color, automated, worn first, with Lotrafilcon B contact lens with color, semi-automated, worn second. Each product worn on a daily wear basis approximately 8 hours a day, 5 days a week, for 2 weeks.
  Interventions: Device: Lotrafilcon B contact lens with color, automated; Device: Lotrafilcon B contact lens with color, semi-automated
- AIR OPTIX® COLORS Semi-auto, then AIR OPTIX® COLORS Auto (Other): Lotrafilcon B contact lens with color, semi-automated, worn first, with Lotrafilcon B contact lens with color, automated, worn second. Each product worn on a daily wear basis approximately 8 hours a day, 5 days a week, for 2 weeks.
  Interventions: Device: Lotrafilcon B contact lens with color, automated; Device: Lotrafilcon B contact lens with color, semi-automated

INTERVENTIONS:
Device: Lotrafilcon B contact lens with color, automated — Silicone hydrogel contact lens with color manufactured via an automated process
  Other Names: AIR OPTIX® COLORS
Device: Lotrafilcon B contact lens with color, semi-automated — Silicone hydrogel contact lens with color manufactured via a semi-automated process
  Other Names: AIR OPTIX® COLORS

SUMMARY:
The purpose of this feasibility study was to compare AIR OPTIX® COLORS contact lenses manufactured using an automated process to AIR OPTIX® COLORS contact lenses manufactured using a semi-automatic process.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign a written Informed Consent form.
* Cylinder ≤ -0.75 diopter (D).
* Able to achieve visual acuity (VA) of at least 20/30 Snellen in each eye at distance with contact lenses (CLCVA) and best corrected visual acuity (BCVA) ≥ 20/25.
* Have spectacles that provide acceptable vision and be willing to wear them if unable to wear the study lenses.
* Successful daily wear of single-vision spherical soft contact lenses in both eyes during the past 3 months for a minimum of 8 hours/day, 5 days/week.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment in this trial.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Currently enrolled in an ophthalmic clinical trial.
* Evidence of systemic or ocular abnormality, infection, or disease likely to affect successful wear of contact lenses or use of accessory solutions, as determined by the investigator.
* Pathologically dry eye.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction | Week 2
  The participant was asked, "Please rate your overall satisfaction based on your experience with the study lenses over the last 2 weeks. When considering your rating, please take into account comfort, vision, and handling, but disregard the appearance of the lenses." Overall satisfaction was rated on a scale of 1-10, with 1=Not at all satisfied, and 10=Completely satisfied.

SECONDARY OUTCOMES:
Overall lens fit | Dispense (Day 0)
  Overall lens fit was assessed by the investigator on a 5-point scale, with +2=Unacceptably loose, +1=Acceptably loose, 0=Optimal, -1=Acceptably tight, -2=Unacceptably tight.
Overall lens fit | Week 2
  Overall lens fit was assessed by the investigator on a 5-point scale, with +2=Unacceptably loose, +1=Acceptably loose, 0=Optimal, -1=Acceptably tight, -2=Unacceptably tight.
Contact Lens Corrected Visual Acuity (CLCVA) | Dispense (Day 0)
  CLCVA (corrected distance monocular visual measurement in normal illumination) was tested for each eye individually while wearing study lenses. Participant read a Snellen chart distant to the participant in normal lighting, with 20/20 Snellen acuity considered normal distance eyesight.
Corrected distance monocular visual measurement in normal illumination reported as Contact Lens Corrected Visual Acuity (CLCVA) | Week 2
  As tested for each eye individually while wearing study lenses. Participant will read a Snellen chart distant to the participant in normal lighting, with 20/20 Snellen acuity considered normal distance eyesight.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Holden Thomas, O.D., Study Director — Alcon Research